CLINICAL TRIAL: NCT00919945
Title: Impact of Early Enteral Feeding on Splanchnic Blood Flow After Surgery for Critical Heart Disease in the Newborn
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Reduced enrollment rate for SV patients due to high competition for studies
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Ben Sivarajan, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000012584
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Congenital Heart Disease
Keywords: Neonates; Congenital Heart Disease; Postoperative Feeding; Splanchnic Blood Flow
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The initial observation period of the study begins in the postoperative period (time 0) after the patient arrives in the Cardiac Critical Care Unit and calibration of the monitors with initial clinically indicated baseline bloodwork is completed. Eligible patients will be randomized when the clinical decision to feed is made (by the treating team) to one of the two treatment arms. Patients in arm 1 will receive continuous nasogastric formula feeding at time 1 and NPO at time 2 (12 hours later).
  Interventions: Other: Continuous feeding at time 1 and NPO at time 2
- 2 (Experimental): The initial observation period of the study begins in the postoperative period (time 0) after the patient arrives in the Cardiac Critical Care Unit and calibration of the monitors with initial clinically indicated baseline bloodwork is completed. Eligible patients will be randomized when the clinical decision to feed is made (by the treating team) to one of the two treatment arms. Patients in arm 2 will receive NPO at time 1 and crossover to continuous nasogastric formula feeding at time 2.
  Interventions: Other: NPO at time 1 and continuous feeding at time 2

INTERVENTIONS:
Other: Continuous feeding at time 1 and NPO at time 2 — Continuous nasogastric formula feeding (using Enfalac with iron 2400 kJ/L at a volume of 1ml/kg/h) at time 1 and NPO at time 2 (12 hours later)
  Arms: 1
Other: NPO at time 1 and continuous feeding at time 2 — NPO at time 1 and continuous nasogastric formula feeding (using Enfalac with iron 2400 kJ/L at a volume of 1ml/kg/h) at time 2 (12 hours later).
  Arms: 2

SUMMARY:
The objective of this study is to determine the impact of early post-operative feeding on splanchnic blood flow, cardiac output and end organ perfusion, and the patients overall clinical outcomes.

DETAILED DESCRIPTION:
Neonates with critical congenital heart disease (CHD) undergoing surgery often have postoperative decreases in cardiac output. These hemodynamic changes can result in varying levels of organ dysfunction, ranging from the subclinical to the more overt. Although this low cardiac output syndrome (LCOS) and accompanying multiorgan dysfunction syndrome (MODS) is in large part transient, the rapidity and completeness of resolution can vary greatly.

During postoperative care in the intensive care unit, knowledge of this phenomenon must be balanced against the desire to initiate enteral nutrition. Many studies have demonstrated that timely initiation of enteral feeds in the intensive care can reduce mortality, morbidity and costs. Practically speaking, the decision to initiate feeds is made based on the patient's postoperative hemodynamic status, a normal lactate, absence of vasopressor agents and presence of bowel sounds. Trophic enteral feeding can usually commence 24h postoperatively, even after complicated neonatal heart surgery,

The vast majority of postoperative neonates suffer no apparent ill effects from this management strategy. However, recent data have demonstrated an exceedingly high incidence (3.3-6.8%) of necrotizing enterocolitis (NEC) in CHD patients; a disease for which diminution in splanchnic blood flow and disruption of the mucosal barrier are felt to play an important role. These data suggest the combination of diminished cardiovascular reserve, cyanosis and increased myocardial oxygen demands may promote the development of NEC.

Preliminary data from Sickkids (Chanthong and Sivarajan, 2008) demonstrates an NEC incidence of 8% in CHD patients. Patients with NEC also accounted for 25% of all cardiac arrests in Cardiac CCU.

ELIGIBILITY:
Inclusion Criteria:

* neonates ≤ 30 days of postnatal age at time of operation
* birthweight > 2.5 kg
* gestational age at birth ≥ 35 weeks
* Patients requiring cardiac surgery who are expected to remain intubated in the CCIU for > 48 hours
* informed consent by parent or guardian
* approval by treating critical care staff physician

Exclusion Criteria:

* patients with heterotaxy or pre-existing renal or abdominal pathology (eg. preoperative diagnosis of NEC).
* need for ECMO after repair within the study period (data up to that point will be recorded and analyzed).
* Parent refusal of formula for purposes of study
* Patient on vasopressin or norepinephrine infusion
* Parent or legal guardian refuse consent

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2009-01; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Change in ultrasound derived bloodflow in superior mesenteric artery after feeding by 1 SD from prefeeding value. | At 0, 6, 12 and 24 hours after arrival at CCU; At 12 and 24 hours after decision to feed is made

SECONDARY OUTCOMES:
Impact of Feeding on: Cardiac Output as measured by continuous mass spectometry, Fractional splanchnic output, Renal Perfusion, Tonometric, Assessment of gastric mucosal pH e. Cerebral oxygen delivery using the NIRS probe | Duration of patient's participation in the study
Correlation and Agreement between: Echo and continuous cardiac output measures; gastric tonometry, SMA PSV and qualitative Bowel Perfusion Index; renal artery PSV and temporal urine output | Duration of patient's participation in the study
Patient Outcomes: Survival, Time to Extubation, Duration of Postop ICU Admission, Duration of Postop hospital Admission, Discharge weight, Number of Nosocomial Infections, Development of NEC | Duration of patient's [articipation in the study

CONTACTS AND LOCATIONS:
Overall Officials: Ben Sivarajan, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada